CLINICAL TRIAL: NCT03944902
Title: Phase 1 Trial of CB-839 in Combination With Niraparib in Platinum Resistant BRCA-wild-type Ovarian Cancer Patients
Brief Title: CB-839 in Combination With Niraparib in Platinum Resistant BRCA -Wild-type Ovarian Cancer Patients
Acronym: BRCA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: will not resume. company choosing not to continue with drug. one participant now off study.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rebecca Arend, Primary Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300002530
Record Dates: First submitted 2019-05-01; First posted 2019-05-10 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Cancer; Resistant BRCA Wild-Type Ovarian Cancer
Keywords: BRCA Wild-Type; Resistant BRCA; Poly (ADP-ribose) polymerase (PARP) Inhibitor Therapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; CB-839

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Dose Escalation using Niraparib and CB-839 (Experimental): The first phase will be a 3+3 design, 3 participants will be enrolled in the first cohort with a fixed dose of Niraparib and CB-839, 600 mg. If there are no dose limiting toxicities (DLT), 3 additional participants will be enrolled in the next cohort (CB-839, 800mg). If 1 of the 3 in the first cohort experiences DLT's, then the additional participants will be enrolled in the same cohort (CB-839, 600mg).
  Interventions: Drug: Cohort 1: Dose Escalation
- Cohort 2: Dose Escalation using Niraparib and CB-839 (Experimental): If there are no DLT's, 3 additional participants will be enrolled in the next cohort with a fixed dose of Niraparib and CB-839, 800mg.
  Interventions: Drug: Cohort 2: Dose Escalation
- Cohort 3: Expansion with Maximum Tolerated Dose (MTD) (Experimental): Patients in this expansion cohort will continue study treatment with the MTD until they experience disease progression, unacceptable toxicity or withdraw consent. Patients who discontinue study treatment for reasons other than Progressive-Free Survival (PFS) will continue to have PFS follow-up visits every 2 months for the first 6 months after treatment, and every 3 months until disease progression, death, or start of another anticancer therapy.
  Interventions: Drug: Cohort 2: Dose Escalation

INTERVENTIONS:
Drug: Cohort 1: Dose Escalation — The first 3 participants will be enrolled on a fixed dose of Niraparib and CB-839, 600mg. Participants will be evaluated for DLT's, if there are none, they will be enrolled in the next cohort.
  Other Names: Niraparib; Zejula; CB-839; Glutaminase inhibitor
  Arms: Cohort 1: Dose Escalation using Niraparib and CB-839
Drug: Cohort 2: Dose Escalation — If no dose limiting toxicities, 3 additional participants will be enrolled in this cohort. Participants will receive a fixed dose of Niraparib and CB-839, 800mg.
  Other Names: Niraparib; Zejula; CB-839; Glutaminase inhibitor
  Arms: Cohort 2: Dose Escalation using Niraparib and CB-839; Cohort 3: Expansion with Maximum Tolerated Dose (MTD)

SUMMARY:
The purpose of this protocol is to investigate the efficacy of the combination of CB-839 with Niraparib in platinum resistant BRCA wild-type ovarian cancer patients. The primary and secondary objectives are to determine the maximum tolerated dose of CB-839 in combination with Niraparib and to determine the response rate and percentage of participants who remain progression free at 6 months.

DETAILED DESCRIPTION:
Based on the scientific rationale, pre-clinical data, and clinical data available to date, and the need for further treatment options in patients that are platinum resistance that are specifically BRCA wild-type. Only patients carrying wild type BRCA genes will be enrolled in the study. The proposed research tests a new therapeutic strategy for ovarian cancer with a very novel mechanistic target: metabolic dependency of ovarian cancer. Pre-clinical results indicate that both serous and clear cells ovarian cancers have upregulation of Hypoxia Inducible Factors (HIF) HIF1a and Hypoxia Inducible Factors (HIF) HIF2a regulated genes. In addition, cell line models of these tumors display sensitivity to CB-839 in vitro. Ovarian cancers resistant to standard platinum chemotherapy may thus respond to treatment with this glutaminase inhibitor. The majority of patients do not present mutations in BRCA or any other genes of the Fanconi pathway, but their tumors may respond to CB-839, which in turn may lead to genomic instabilities due to nucleotide deprivation; therefore, CB-839 could sensitize the tumors to treatment with Niraparib.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Estimated life expectancy of at least 3 months
* Measurable disease; at least one tumor lesion/lymph node that meets the RECIST 1.1 criteria for measurability
* Negative serum or urine pregnancy test within 3 days prior to the first dose
* Serum creatinine <= 2.0 x upper limit of normal (ULN)
* Adequate hematological function
* Alanine aminotransferase (ALT) & aspartate aminotransferase (AST) <3.0 x ULN
* Total bilirubin <=1.5 x ULN

Exclusion Criteria:

* Prior treatment with CB-839 or a PARP inhibitor
* Receipt of any anticancer therapy within the following windows:
* Small molecule tyrosine kinase inhibitor therapy (including investigational) within 2 weeks or 5 half-lives, whichever is longer
* Any type of anti-cancer antibody within 4 weeks
* Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before randomization
* Subjects with clinically relevant ongoing complications from prior radiation therapy
* Other investigational therapy within 2 weeks or 5 half-lives, whichever is longer
* Any other current or previous malignancy within he past three years except:
* Adequately treated basal cell or squamous cell skin cancer
* Carcinoma in situ of the cervix
* Prostate cancer with stable prostate specific antigen (PSA) levels for >3 years
* Other neoplasm that, in the opinion of the Principal Investigator, will not interfere with the study-specific endpoints

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Access toxicity as evidenced by the number and percent of treatment adverse events. | Baseline through Week 1
  Any CTCAE v4.0 grade 3 except with some identified exceptions: Grade 3-4 nausea, vomiting and diarrhea, Grade 3 transaminitis present for <= 7 days, Grade 3 laboratory abnormalities (correctable & asymptomatic), Grade 3 ALT or AST elevation, Grade 3 thrombocytopenia or neutropenia, and Grade 4 anemia.
Access toxicity as evidenced by the number and percent of treatment adverse events. | Baseline through Week 2
  Any CTCAE v4.0 grade 3 except with some identified exceptions: Grade 3-4 nausea, vomiting and diarrhea, Grade 3 transaminitis present for <= 7 days, Grade 3 laboratory abnormalities (correctable & asymptomatic), Grade 3 ALT or AST elevation, Grade 3 thrombocytopenia or neutropenia, and Grade 4 anemia.
Access toxicity as evidenced by the number and percent of treatment adverse events. | Baseline through Week 3
  Any CTCAE v4.0 grade 3 except with some identified exceptions: Grade 3-4 nausea, vomiting and diarrhea, Grade 3 transaminitis present for <= 7 days, Grade 3 laboratory abnormalities (correctable & asymptomatic), Grade 3 ALT or AST elevation, Grade 3 thrombocytopenia or neutropenia, and Grade 4 anemia.
Access toxicity as evidenced by the number and percent of treatment adverse events. | Baseline through Week 4
  Any CTCAE v4.0 grade 3 except with some identified exceptions: Grade 3-4 nausea, vomiting and diarrhea, Grade 3 transaminitis present for <= 7 days, Grade 3 laboratory abnormalities (correctable & asymptomatic), Grade 3 ALT or AST elevation, Grade 3 thrombocytopenia or neutropenia, and Grade 4 anemia.
Access toxicity as evidenced by the number and percent of treatment adverse events. | Baseline through Week 12
  Any CTCAE v4.0 grade 3 except with some identified exceptions: Grade 3-4 nausea, vomiting and diarrhea, Grade 3 transaminitis present for <= 7 days, Grade 3 laboratory abnormalities (correctable & asymptomatic), Grade 3 ALT or AST elevation, Grade 3 thrombocytopenia or neutropenia, and Grade 4 anemia.
Access toxicity as evidenced by the number and percent of treatment adverse events. | Baseline through Week 24
  Any CTCAE v4.0 grade 3 except with some identified exceptions: Grade 3-4 nausea, vomiting and diarrhea, Grade 3 transaminitis present for <= 7 days, Grade 3 laboratory abnormalities (correctable & asymptomatic), Grade 3 ALT or AST elevation, Grade 3 thrombocytopenia or neutropenia, and Grade 4 anemia.
Access toxicity as evidenced by the number and percent of treatment adverse events. | Baseline through Week 48
  Any CTCAE v4.0 grade 3 except with some identified exceptions: Grade 3-4 nausea, vomiting and diarrhea, Grade 3 transaminitis present for <= 7 days, Grade 3 laboratory abnormalities (correctable & asymptomatic), Grade 3 ALT or AST elevation, Grade 3 thrombocytopenia or neutropenia, and Grade 4 anemia.

SECONDARY OUTCOMES:
Determine the response rate by the percentage of patients that remain progression free as measured by the Response Evaluation Criteria in Solid Tumors (RECIST). | Baseline through 6 months
  Response will be evaluated by the revised RECIST. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes. Assessment of association among biomarkers will be carried out by dose level and cycle.
Determine progression rate by the percentage of patients that have disease progression as measured by the Response Evaluation Criteria in Solid Tumors (RECIST). | Baseline through 6 months
  Progression will be evaluated by the revised RECIST. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes. Assessment of association among biomarkers will be carried out by dose level and cycle.
Determine the response rate by the percentage of patients that remain progression free as measured by the Response Evaluation Criteria in Solid Tumors (RECIST). | Baseline through 12 months
  Response will be evaluated by the revised RECIST. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes. Assessment of association among biomarkers will be carried out by dose level and cycle.
Determine the progression rate by the percentage of patients that have disease progression as measured by the Response Evaluation Criteria in Solid Tumors (RECIST). | Baseline through 12 months
  Progression will be evaluated by the revised RECIST. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes. Assessment of association among biomarkers will be carried out by dose level and cycle.
Determine the response rate by the percentage of patients that remain progression free as measured by the Response Evaluation Criteria in Solid Tumors (RECIST). | Baseline through 18 months
  Response will be evaluated by the revised RECIST. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes. Assessment of association among biomarkers will be carried out by dose level and cycle.
Determine the progression rate by the percentage of patients that have disease progression as measured by the Response Evaluation Criteria in Solid Tumors (RECIST). | Baseline through 18 months
  Progression will be evaluated by the revised RECIST. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes. Assessment of association among biomarkers will be carried out by dose level and cycle.
Determine the response rate by the percentage of patients that remain progression free as measured by the Response Evaluation Criteria in Solid Tumors (RECIST). | Baseline through 24 months
  Response will be evaluated by the revised RECIST. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes. Assessment of association among biomarkers will be carried out by dose level and cycle.
Determine the progression rate by the percentage of patients that have disease progression as measured by the Response Evaluation Criteria in Solid Tumors (RECIST). | Baseline through 24 months
  Progression will be evaluated by the revised RECIST. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes. Assessment of association among biomarkers will be carried out by dose level and cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Arend, MD, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCSF, San Francisco, California
  - MAYO Clinic, Rochester, Minnesota
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
To be determined.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The above documents will be posted on CT.gov and available as long as study record is posted.
Access Criteria: To be determined.